CLINICAL TRIAL: NCT07250724
Title: A Prospective, Observational Study to Evaluate C. Difficile Toxin Levels in Stool in Healthy Individuals Following Standard of Care Antibiotic Treatment for CDI.
Brief Title: C. Difficile Toxin Levels in Stool From Healthy Individuals Following Standard of Care Antibiotic Treatment for CDI.
Status: Recruiting | Type: Observational
Sponsor: Bactolife A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: AFCRO-193
Record Dates: First submitted 2025-09-26; First posted 2025-11-26 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Clostridioides Difficile Infection Recurrence
Keywords: C. Diff; Clostridioides Difficile; Clostridioides Difficile Infection; Clostridioides Difficile Infection Recurrence; Clostridioides Difficile Recurrence; C. Diff recurrence
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples. DNA sequencing plenned, but only to look at bacterial DNA, not human DNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Participants that are undergoing standard of care antibiotic treatment for their second C. Diff infection will be followed for 8 weeks after completing antibiotic treatment. — Participants that are undergoing standard of care antibiotic treatment for their second C. Diff infection will be followed for 8 weeks after completing antibiotic treatment.

SUMMARY:
Hospitals and clinics interested in participating in this multi-site study, please contact the people mentioned under "Contacts and Locations".

The goal of this study is to map the risk of having a C. Difficile infection recurrence (rCDI) after being treated with standard-of-care antibiotics for a C. Difficile infection.

The main questions it aims to answer are:

* What is the recurrence rate of CDI in the 8 weeks following antibiotic treatment for a first recurrence of CDI?
* Does toxin levels of Toxin A and/or B from C. Diff. at baseline predict CDI recurrence risk?

Participants will:

* Undergo standard of care Antibiotic treatment for first recurrence of CDI
* Visit their clinic at 4 different visits over a time period of approximately 9 weeks. (Visits can also be performed remote/via phone call.)

DETAILED DESCRIPTION:
Hospitals and clinics interested in participating in this multi-site study, please contact the people mentioned under "Contacts and Locations".

This prospective observational study will enrol 60 otherwise healthy adults with a documented history of first recurrent Clostridioides difficile infection (rCDI). Eligible participants must have had a confirmed positive toxin B test for C. difficile, with the initial infection occurring within the past 12 months. At the time of enrolment (Day 0), participants must have completed a standard-of-care oral antibiotic therapy for their first rCDI no more than five days prior and be asymptomatic for CDI. Potential participants will sign an informed consent form at their initial visit to their doctor (visit 1) and provide a stool sample for c diff testing. Participants will only be considered 'enrolled' if their stool sample is positive for toxin B and they meet all other criteria at visit 2 (week 0).

The primary objective of the study is to measure the rate of CDI recurrence within an 8-week follow-up period. The secondary objective is to assess stool levels of Toxin A and B at baseline, week 2, and week 8. The second objective will enable exploration of the reliability of using high-sensitivity assays for toxin detection in stool. Further, potential correlations between post-treatment stool toxin levels and rCDI development will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide signed and dated informed consent
* Males and females between 18 - 75 years old inclusive
* Documented history of first recurrent Clostridioides difficile (former Clostridium difficile) infection (rCDI), confirmed by a positive C. difficile test (Toxin A+B positive or Toxin B only), with initial infection occurring within the previous 12-months.
* Must, in accordance with standard of care practices, have completed a SOC oral antibiotic therapy for the first rCDI no more than 5 days prior to the date of enrolment (baseline visit- Day 0).
* Must not have any CDI-related symptoms when enrolled in the study at baseline (Day 0).

Exclusion Criteria:

* Current episode of CDI or delayed symptom resolution from previous recurrence, according to the physical exam and investigator assessment
* Toxin A positive, and Toxin B negative C. difficile test.
* Planned CDI recurrence treatment for the duration of the study e.g., fecal microbiome transplant, probiotics, Live Biotherapeutic Products (LBPs)
* Those who are on further antibiotic treatment following initial rCDI antibiotic therapy completion.
* Pregnant or lactating women or women who intend to become pregnant within the next 3 months.
* Subjects presenting with active diarrhoea (3 or more stools per 24-hour period) and within Bristol stool scale range of 5-7 at baseline.
* Has any significant acute or chronic coexisting health conditions that would prevent them from fulfilling the study requirements, put the Participant at risk or would confound the interpretation of the study results as judged by the investigator on the basis of medical history and routine laboratory test results.

  * Ostomized participants, parenteral nutrition users
  * Patients with active Pancreatitis
  * Active, non-controlled intestinal diseases such as IBS, IBD, Crohn's Disease, ulcerative colitis, celiac disease, or other chronic diarrheal illness
* Currently or recently taking a medication that the investigator believes would interfere with the objectives of the study or pose a safety risk or confound the interpretation of the study results.
* Individuals who, in the opinion of the investigator, are considered to be poor attendees or unlikely for any reason to be able to comply with the study.
* Participants may not be participating in other clinical studies. If the participant has previously taken part in an experimental study, the Investigator must ensure sufficient time has elapsed before entry to this study to ensure the integrity of the results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective observational study will enrol 60 otherwise healthy adults with a documented history of first recurrent Clostridioides difficile infection (rCDI). Eligible participants must have had a confirmed positive toxin B test for C. difficile, with the initial infection occurring within the past 12 months. At the time of enrolment (Day 0), participants must have completed a standard-of-care oral antibiotic therapy for their first rCDI no more than five days prior and be asymptomatic for CDI. Potential participants will sign an informed consent form at their initial visit to their doctor (visit 1) and provide a stool sample for c diff testing. Participants will only be considered 'enrolled' if their stool sample is positive for toxin B and they meet all criteria at visit 2.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects experiencing CDI recurrence in the time period between baseline and end of study follow-up. | Within the 8 week time period between baseline and end of follow-up
  CDI recurrence will be defined as the development of a new episode of diarrhoea (3 or more loose stools in 24 or fewer hours) associated with a positive stool test for toxigenic C. difficile following clinical cure of the initial CDI episode.

CONTACTS AND LOCATIONS:
Overall Officials: Brynjulf Mortensen, pHD, Study Director — Bactolife A/S
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No